CLINICAL TRIAL: NCT04309149
Title: Market Research - Acceptability Study for a Range of New MCT Based Products (Dr Schär - Kanso MCT) Kanso MCT 100% Oil Kanso MCT 77% Oil Kanso MCT 83% Margarine
Brief Title: Market Research - Acceptability Study for a Range of MCT Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Schär AG / SPA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Kanso 1
Record Dates: First submitted 2020-03-09; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Ketosis; Epilepsy; Ketogenic Diet; Fatty Acid Oxidation Disorder; Malabsorption
MeSH Terms: conditions — Ketosis; Epilepsy; Malabsorption Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MCT fats (Experimental): Kanso MCT oils and margarine will be consumed daily for 7 days each to assess tolerability and compliance
  Interventions: Dietary Supplement: MCT fats

INTERVENTIONS:
Dietary Supplement: MCT fats — Subjects will be asked to take 3 new MCT products for 7 days each over a 25 day period (21 days taking the new products with 2 days between each new product trialled).

SUMMARY:
This is a market research, observational study to evaluate the tolerability and acceptability of MCT supplements for young children and young people with intractable epilepsy, GLUT-1 or PDHD from 3 years to adulthood. Patients with a confirmed diagnosis of a fatty acid oxidation disorder, which requires a specialist diet including MCT will be included in this study

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of epilepsy or a fatty acid oxidation disorder requiring a ketogenic or a specialist diet as part of their treatment, which includes MCT.
* Subjects who are new to or already taking an MCT oil and are willing to try each of the 3 study products for 7 days each. 21 days taking product with 2 days between new product trialled.
* Patients aged 3 years of age to adulthood.
* Written informed consent obtained from patient or parental caregiver.

Exclusion Criteria:

* Presence of serious concurrent illness
* Investigator's uncertainty about the willingness or ability of the patient to comply with the protocol requirements
* Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study.
* Any patients having taken antibiotics over the previous 2 weeks leading up to the study.
* Patients less than 3 years of age.

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal tolerance | 7 days for each product, maximum 25 days
  Questionnaire detailing any GI symptoms, severity and change from usual The collection of daily data about the gastrointestinal tolerance of the product
Product compliance | 7 days for each product, maximum 25 days
  Daily questionnaire on amounts offered and amounts actually consumed, compared to recommended amount.
Product palatability | 7 days for each product, maximum 25 days
  Questionnaire data captured to evaluate taste
Product acceptability | 7 days for each product, maximum 25 days
  Brief tick-box questionnaire on overall liking and acceptability of product

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Bristol Royal Hospital for Children, Bristol
  - Royal Manchester Children's Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No
This study will be used to demonstrate acceptability for registration and reimbursement of these foods for special medical purposes.